CLINICAL TRIAL: NCT07107490
Title: AN OPEN-LABEL, MULTICENTER PHASE I STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND PRELIMINARY ANTI-TUMOR ACTIVITY OF ALPS12 IN PATIENTS WITH EXTENSIVE STAGE SMALL CELL LUNG CANCER
Brief Title: A PHASE I STUDY OF ALPS12 IN PATIENTS WITH EXTENSIVE STAGE SMALL CELL LUNG CANCER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALP102CT
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation part (Experimental): Patients will receive ALPS12 as a single agent following pretreatment of obinutuzumab to determine the MTD by evaluating DLTs in patients with extensive stage small cell lung cancer.
  Interventions: Drug: ALPS12; Drug: obinutuzumab
- Expansion part (Experimental): Patients will receive ALPS12 as a single agent following pretreatment of obinutuzumab to evaluate the antitumor effect.
  Interventions: Drug: ALPS12; Drug: obinutuzumab

INTERVENTIONS:
Drug: ALPS12 — ALPS12 as an IV infusion
Drug: obinutuzumab — Obinutuzumab as an IV infusion

SUMMARY:
This study is a phase I, open-label, multicenter trial designed to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and antitumor activity of ALPS12 in patients with extensive-stage small cell lung cancer. The study consists of two parts: a dose-escalation part and an expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years at time of informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Histologically documented extensive stage small cell lung cancer
* Disease recurrence documented after at least one prior systemic therapy.
* Confirmed availability of representative archival tumor specimens or fresh tumor specimen.
* Measurable disease per RECIST v.1.1.
* Adequate hematologic and end organ function

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or breastfeeding during the study
* History or complication of clinically significant autoimmune disease
* a positive HIV antibody test at screening
* Active hepatitis B or hepatitis C
* Prior treatment with anti-CD137 antibody drugs, anti-CD3 antibody drugs, and/or DLL3-targeted therapies
* Patients who have received any investigational or approved anticancer therapy, including hormone therapy and/or radiotherapy, within 21 days prior to the first administration of the investigational drug.
* History of Grade 4 immune-related adverse events caused by prior anti-PD-L1/PD-1 antibody drugs or anti-CTLA-4 antibody drugs (excluding asymptomatic elevations in serum amylase/lipase)
* Patients who discontinued immunotherapy due to Grade 3 immune-related adverse events caused by prior anti-PD-L1/PD-1 antibody drugs or anti-CTLA-4 antibody drugs (excluding asymptomatic elevations in serum amylase/lipase), and/or patients who experienced Grade 3 immune-related adverse events caused by immunotherapy within 6 months prior to the first administration of the investigational drug
* Patients who received a live attenuated vaccine within 4 weeks prior to the first administration of the investigational drug
* History or clinical evidence of primary central nervous system (CNS) malignancy, symptomatic CNS metastases, CNS metastases requiring any anti tumor treatment, or leptomeningeal disease
* Current or past CNS diseases (e.g., stroke, epilepsy, CNS vasculitis, neurodegenerative diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
All part : Adverse events of ALPS12[safety and tolerability] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Incidence, nature, and severity of AEs graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0, and CRS and Immune effector cell-associated neurotoxicity syndrome (ICANS) graded according to the ASTCT Consensus Grading Criteria
Dose Escalation part : Dose-limiting toxicities (DLTs) and PK profile of ALPS12[safety and tolerability] | From Cycle 1 Day 1 to the administration of ALPS12 on Cycle 2 Day 1 (Cycle 1 is 21 days)
  Nature and frequency of DLTs, AEs, PK and PD profiles
Dose Escalation part : Immunogenicity of ALPS12 | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Incidence of ADAs to ALPS12 and potential correlation with PK parameters and safety
Expansion part : Preliminary anti-tumor activity of ALPS12 when administered at selected dose(s) based on tumor assessment in patients with extensive stage SCLC | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Objective response, defined as a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, as determined by the Investigators

SECONDARY OUTCOMES:
Objective response rate(ORR)[preliminary efficacy] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  ORR assessed per RECIST v.1.1 by the investigators.
Disease control [preliminary efficacy] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  defined as the proportion of patients who have CR, PR, or stable disease (SD) as best overall response per RECIST v.1.1 as determined by the investigator.
Duration of response (DoR)[preliminary efficacy] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Duration of response (DoR), defined as the time from the first occurrence of CR or PR to progression disease (PD) or death from any cause (whichever occurs first), per the investigator according to RECIST v.1.1
Progression-free survival (PFS)[preliminary efficacy] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Progression-free survival (PFS), defined as the time from administration of first study treatment to the first occurrence of disease progression or death from any cause, as determined by the investigator according to RECIST v.1.1
Overall survival (OS)[preliminary efficacy] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Overall survival (OS), defined as the time from administration of first study treatment to death from any cause
Immunogenicity of obinutuzumab | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Incidence of ADAs to obinutuzumab and potential correlation with PK parameters and safety
Maximum serum concentration (Cmax) and Area under the concentration time-curve (AUC) of ALPS12 with obinutuzumab[PK profile] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Serum ALPS12 concentration and its PK parameters including Cmax and AUC etc.
Adverse events of obinutuzumab[safety and tolerability] | From screening until study completion or treatment discontinuation, assessed up to the end of the study (approximate 42 months)
  Incidence, nature, and severity of adverse events graded according to NCI Common Terminology CTCAE v5.0, with severity of CRS determined according to the American Society for Transplantation and Cell Therapy (ASTCT) Consensus Grading Criteria(In parts with obinutuzumab premedication)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co.Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (6):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Kindai University Hospital, Sakai, Osaka
  - Niigata Cancer Center Hospital, Niigata
- Show Chwan Memorial Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).